CLINICAL TRIAL: NCT03001336
Title: Association Between Thyroid Function and Diabetes Complications in Elderly Patients With Type 2 Diabetes Mellitus in China
Brief Title: Thyroid Function and Diabetes Complications
Status: Completed | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: DIA-THY-1
Record Dates: First submitted 2016-12-12; First posted 2016-12-23 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2011-01

CONDITIONS: Diabetes; Thyroid Disease
Keywords: Thyroid; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus; Thyroid Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: no intervention — This is a cross-sectional study

SUMMARY:
The purpose of this study is to investigate the potential association between thyroid function and diabetes complications in the elderly subjects with type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
Aims: We investigated the potential association between thyroid parameters and microalbuminuria in the euthyroid elderly subjects with type 2 diabetes mellitus (T2DM).

Subjects: Elderly inhospital patients with T2DM who visited in the Department of Endocrinology at the Nanjing First Hospital from January 2011 to December 2012.

Methods: Clinical factors, serum levels of glucose, lipids, free triiodothyronine (FT3), free thyroxine (FT4), thyroid-stimulating hormone (TSH), thyroid autoantibodies,24h urine albuminuria and fluorescence fundus angiography are conducted.

The relationships levels of thyroid function and diabetic complications are analysed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are ≥ 60 years old, with T2DM and the diagnostic criteria of T2DM is according to the World Health Organization in 1999.
2. Patients have normal thyroid function and negative for thyroid autoantibodies, such as thyroid peroxidase antibody (TPOAb) or thyroglobulin antibody (TGAb).

Exclusion Criteria:

1. Patients with a history of thyroid disease or chronic liver disease or nondiabetic renal problems or cancer.
2. Patients use systemic drug therapy such as thyroxine, anti-thyroid drugs, glucocorticoids and oral contraceptives.
3. Patients are pregnant or lactating women.
4. Patients with acute intercurrent illness of diabetes.
5. Patients with an acute infection.
6. Patients with a history of drug abuse alcohol dependence in the past 5 years.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes who visited in the Department of Endocrinology at the Nanjing First Hospital from January 2011 to December 2012 were enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Diabetic retinopathy which is diagnosed by the measurement of fundus fluorescein angiography. (Diabetic retinopathy is clinically graded based on the international clinical diabetic retinopathy severity scales.) | Day One

SECONDARY OUTCOMES:
24h-albuminuria | Day One

IPD SHARING:
Plan to Share IPD: No